CLINICAL TRIAL: NCT03974048
Title: Identification of the Epigenetic Response to Trauma - a Prospective, Observational Study
Brief Title: Identification of the Epigenetic Response to Trauma
Acronym: TrauMeth
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Trine Grodum Eskesen, Medical Doctor, Rigshospitalet, Denmark
Other Study IDs: VD-2019-161
Record Dates: First submitted 2019-05-29; First posted 2019-06-04 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Trauma; Injuries
Keywords: Epigenetics; DNA methylation; Trauma
MeSH Terms: conditions — Wounds and Injuries | interventions — Blood Specimen Collection; DNA Methylation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples are obtained from patients to investigate DNA methylation profiles
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trauma patients: All trauma patients admitted to Rigshospitalet's trauma center will have a blood sample taken during the initial treatment and 30 days after the trauma.
  Interventions: Diagnostic Test: Blood samples for DNA methylation analysis
- Patients admitted for elective orthopedic surgery: The patients will have a blood sample taken before and after surgery and again 30 days after the surgery.
  Interventions: Diagnostic Test: Blood samples for DNA methylation analysis

INTERVENTIONS:
Diagnostic Test: Blood samples for DNA methylation analysis — DNA from blood samples will be isolated and analyzed for genome-wide DNA methylation patterns using the Infinium HumanMethylationEPIC BeadChip (Illumina, San Diego, CA, USA).

SUMMARY:
The objective of this study is to investigate potential early alterations in the DNA methylation profile after severe trauma and to investigate if the early marks persist.

DETAILED DESCRIPTION:
Background: Severe trauma is an extreme physical exposure, which may have significant consequences for the patient. In addition to anatomical injury and hemodynamic compromise, severe trauma causes an immense and rapid systemic immune reaction. At the genomic level, trauma has been found to significantly increase gene expression in circulating leukocytes, and preliminary data is also emerging that trauma may even cause epigenetic (DNA methylation) alterations.

Epigenetics, including DNA methylation, have been suggested as a mediator of genetic risk and to play a significant role in subsequent non-traumatic disease. Within the field of trauma DNA methylation has only been sparsely studied, but a few studies of traumatized animals have suggested that DNA methylation alterations may occur in relation to trauma. Even though DNA methylation is highly dynamic, some marks have been found to be stable over time, and thus may have long-term consequences.

An increasing understanding of the role of epigenetics in disease development and response may pave the way for new treatment targets and modalities for multiple diseases including trauma.

Research question: Does trauma induce immediate (<4 hours) and persistent (30 days post-trauma) changes in the epigenome of peripheral blood cells, and do epigenetic changes correlate with patient recovery?

Objectives: To identify potential early alterations in the DNA methylation profile after severe trauma AND to investigate if the early marks persist.

Study design: A prospective, observational, cohort study of trauma patients admitted to RH's trauma center. The trauma cohort will be compared to a cohort of patients admitted for elective orthopedic surgery in terms of DNA methylation profile in blood cells pre-trauma/surgery, immediately post-trauma/surgery, and 30-45 days post-trauma/surgery.

DNA methylation profiles will be assessed by array technique using Illumina's MethylationEPIC Bead-Chip.

Primary outcome: Immediate (<4 hours) post-trauma DNA methylation profile in blood cells.

Secondary outcomes: Pre-trauma/surgery DNA methylation profile, change in DNA methylation from pre-trauma/surgery to immediately and 30 days post-trauma/surgery, occurrence of organ dysfunction, sepsis, septic shock, 30-day mortality, ICU admission > 24 hours, ICU length of stay (LOS), hospital LOS.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Trauma patients: Admitted to Rigshospitalet's trauma center generating a trauma team activation.
* Surgical controls: Admitted for elective surgery (non-traumatic cause) at the orthopedics department AND

  * Only one surgical procedure planned from study day 0 to study day 45.
  * Expected procedure length of at least 60 minutes.

Exclusion Criteria:

* Not able to obtain informed consent and not possible to obtain consent from a next-of-kin.
* Trauma patients:

  * Secondary transfers.
  * Pre-hospital blood transfusion OR blood transfusion in the trauma center before the first blood sample is obtained.
  * First blood sample taken later than 4 hours after the trauma.
  * Patients in cardiac arrest before/after hospital admission.
  * Additional traumatic exposure requiring hospital admission between the collection of the primary blood sample and the follow-up blood sample (will cause exclusion from follow-up blood sample).
  * Surgery not related to the trauma between the collection of the primary blood sample and the follow-up blood sample (will cause exclusion from follow-up blood sample).
* Surgical controls:

  * Surgical procedures due to cancer or fractures.
  * Traumatic exposure requiring hospital admission between the collection of the primary blood sample and the follow-up blood sample (will cause exclusion from follow-up blood sample).
  * Additional, unplanned surgery between the collection of the primary blood sample and the follow-up blood sample (will cause exclusion from follow-up blood sample).
  * First post-operative blood sample taken later than 4 hours after surgical end time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of all trauma patients admitted to RH's trauma center generating a trauma team activation.
  The control group will consist of patients admitted to RH's orthopedic department for elective surgery.
Sampling Method: Probability Sample
Enrollment: 365 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Immediate DNA methylation profile | Day of trauma/surgery
  Immediate (< 4 hours) post-trauma DNA methylation profile in blood cells compared to the pre-surgery (baseline) and immediate post-surgery (< 4 hours) DNA methylation profile in blood cells.

SECONDARY OUTCOMES:
Pre-trauma/-surgery DNA methylation profile | Pre-trauma/surgery
  Pre-trauma (if possible to obtain from an existing biobank) DNA methylation profile in blood cells compared to pre-surgery.
Stability of DNA methylation profile | 30-45 days after trauma/surgery
  Persistence of the DNA methylation profile in blood cells 30-45 days after the trauma compared to surgical patients.
Change in DNA methylation profile; pre-trauma/-surgery to post-trauma/-surgery | Day of trauma/surgery
  Change in DNA methylation profile in blood cells from pre-trauma (if possible to obtain) to immediately post-trauma compared to surgical patients.
Change in DNA methylation profile; immediately post-trauma/-surgery to one month post-trauma/-surgery | 0 to 30-45 days after trauma/surgery
  Change in DNA methylation profile in blood cells from immediately post-trauma to 30-45 days post-trauma compared to surgical patients.
DNA methylation changes in relation to injury severity | Day 0-45 after trauma/surgery
  Association of DNA methylation changes with injury severity. This will be done by comparing the DNA methylation profiles among patient with an injury severity score (ISS) < 15 and patients with an ISS > 15.
Organ dysfunction | Day 30 after trauma/surgery
  Occurrence of organ dysfunction (increase of ≥ 2 in SOFA-score)
Sepsis/septic shock | Day 30 after trauma/surgery
  Occurrence of sepsis or septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Steinmetz, MD, Ph.D., Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No